CLINICAL TRIAL: NCT02139345
Title: A Prospective, Randomized, Multicenter Clinical Study to Compare the Safety and Efficacy of TC-A PS Total Knee System With TC-PLUS Solution PS Total Knee System in Chinese Subjects
Brief Title: TC-A Registration Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew Medical (Shanghai) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-4060-04
Record Dates: First submitted 2014-05-07; First posted 2014-05-15 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Primary Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Avascular Necrosis
Keywords: Osteoarthritis; Rheumatoid arthritis; Post-traumatic arthritis; Avascular necrosis; AVN
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteonecrosis; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Subject was randomized to receive the treatment of investigational device or the comparator.
Who Masked: Outcomes Assessor
Masking Description: Investigator who assesses KSS score is blinded to the subject's treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TC-A PS (Experimental): Subject will be implanted with the TC-A PS Total Knee Replacement System
  Interventions: Device: TC-A PS Total Knee Replacement System
- TC-PLUS Solution PS (Active Comparator): Subject will be implanted with the TC-PLUS Solution PS Total Knee Replacement System.
  Interventions: Device: TC-PLUS Solution PS Total Knee Replacement System

INTERVENTIONS:
Device: TC-A PS Total Knee Replacement System — Subject will be implanted with the TC-A PS Total Knee Replacement System
  Other Names: TC-A PS
  Arms: TC-A PS
Device: TC-PLUS Solution PS Total Knee Replacement System — Subject will be implanted with the TC-PLUS Solution PS Total Knee Replacement System
  Other Names: TC-PLUS Solution PS
  Arms: TC-PLUS Solution PS

SUMMARY:
This is a prospective, randomized, multicenter clinical study to compare the safety and efficacy of TC-A PS total knee system with TC-PLUS Solution PS total knee system in Chinese subjects.

DETAILED DESCRIPTION:
Osteoarthritis (OA), also known as degenerative joint disease or hyperostosis, is the most common cause of knee arthritis. Pain, dyskinesia and disability induced by osteoarthritis impact severely on the subject's health and quality of life. Knee osteoarthritis is very common in the elderly population. As life expectancy has increased, the incidence of osteoarthritis rose significantly during the 20th century. For people over 60 years of age, approximately 50% show signs of osteoarthritis on x-rays, among which 35% -50% show clinical signs. For people over the age of 75, 80% had osteoarthritis symptoms.

There has been an increase in imported knee prostheses during the past decade, so that surgeons now have more choices of implants. However, the high cost of imported prostheses has become a barrier to the development of TKA in China and caused many OA subjects requiring immediate TKA to have to delay or miss their surgery. The development and promotion of high-quality domestic joint implants and surgical instruments is the key to the development of TKA technique in China.

The primary objective of this study is to demonstrate non-inferiority of subjects implanted with the TC-A PS total knee system compared to a randomized concurrent control group of subjects implanted with the TC-PLUS Solution PS total knee system in terms of Knee Society Clinical Score (KSCS) at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 50 and 75 years inclusive of Chinese ethnicity.
* Subject presents with primary osteoarthritis, rheumatoid arthritis, post-traumatic arthritis or avascular necrosis of knee joint requiring primary total knee replacement with the PS knee system.
* Subject who is able to give voluntary, written informed consent to participate in the study and from whom consent has been obtained by signing and dating an EC-approved consent form.
* Subject who is able to understand this clinical study, co-operates with the investigational procedures and is willing to return to the hospital for all the required post-operative follow-ups for up to 12 months.
* Life expectancy of subject is over 2 years.

Exclusion Criteria:

* Bilateral knee disease with the anticipated need for bilateral knee implant during study participation (i.e., within the next 12 months).
* Subject has known or suspected metal sensitivity.
* Subject is known to have insufficient femoral or tibial bone stock resulting from conditions such as cancer, distal femoral/proximal tibial osteotomy, significant osteoporosis or metabolic bone disorders, which cannot provide adequate support and/or fixation to the prosthesis.
* Subject is severely obese (BMI>35).
* Subject has hip arthritis and/or replacement.
* Subject had an active infection or sepsis (treated or untreated)
* Subject has conditions that may compromise implant stability or postoperative recovery (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
* Subject has an emotional or neurological condition that would affect their ability or willingness to participate in the study (e.g. mental illness, mental retardation).
* Subject is immunosuppressed, has an autoimmune disorder, or an immunosuppressive disorder. For examples, subject is on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses) or has acquired immunodeficiency syndrome (AIDS).
* Subject is a woman who is pregnant or lactating，or intends to become pregnant during the course of the study.
* Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits.
* Subject was enrolled in another investigational drug, biologic, or device study in the last 12 months.
* Known alcohol and/or drug abuse

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
The Original Knee Society Clinical Score (KSCS) | 1 year post-operative
  The Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. For the results, a score of 80-100 = excellent, 70-79 = good; 60-69 = fair; and < 60 = poor.

SECONDARY OUTCOMES:
The Original Knee Society Functional Score (KSFS) | 1 year post-operative
  The Knee Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. For the result, a score of 80-100 = excellent, 70-79 = good; 60-69 = fair; and < 60 = poor.
Revision for any reason | Up to 1 year post-operative
  Revision for any reason will be assessed and documented up to 1 year post-operative.
Linear radiolucencies and radiographic abnormalities | Up to 1 year post-operative
  Radiographic measurements will be taken of linear radiolucencies and the radiographs will be evaluated for any abnormalities.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 1 year post-operative
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of subjects with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties.
SF-12 Health Survey | 1 year post-operative
  The SF-12 Health Survey was first developed in 1995 as a shorter version of the SF-36 Health Survey used for measuring the overall health condition of the general population. The usefulness of SF-12 is improved by its simplicity and less time needed for completion, and it has a good reliability on the evaluation of quality of life. The SF-12v2 Health Survey is a 12-item generic Health-Related Quality of Life measure consisted of eight subscales: Physical functioning (PF), Role physical (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Role emotional (RE) and Mental health (MH); and two composite summary scores: Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. All subscales and summary scores were ranged from 0-100. The higher the SF-12 score, the better the HRQOL outcome.
Number of subjects with adverse events | Up to 1 year post-operative
  Safety will be evaluated by collecting the frequency and nature of all postoperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, Professor, Principal Investigator — Peking University People's Hospital
Locations (4):
- China (4):
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Peking University People's Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No